CLINICAL TRIAL: NCT06957665
Title: Treatment Outcomes of Temporomandibular Disorders Using Stabilization Splint Supported by the T-scan System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, DUC NGUYEN MINH, Lecturer, Hanoi Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHMCK62722815
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2023-06

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: Temporomandibular Disorders; Stabilization Splints; T-scan System
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Intervention Model Description: A single-group, non-randomized clinical study where all enrolled participants received stabilization splint therapy supported by T-scan system-assisted occlusal adjustment. No control or comparison group was used.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stabilization Splint with T-scan Assisted Adjustment (Experimental): Participants received a custom-fabricated stabilization splint (Michigan splint) with occlusal adjustments guided by the T-scan system. The splints were adjusted based on both articulating paper and real-time occlusal force analysis provided by the T-scan system to optimize occlusal balance. No control or comparator arm was used.
  Interventions: Device: T-scan Assisted Occlusal Adjustment with Stabilization Splint

INTERVENTIONS:
Device: T-scan Assisted Occlusal Adjustment with Stabilization Splint — Participants were treated with a custom-fabricated stabilization splint (Michigan-type) whose occlusion was adjusted using the T-scan system (Tekscan, Norwood, MA, USA) to measure and optimize occlusal force distribution. The T-scan system was used in conjunction with articulating paper to guide occlusal refinement until bilateral force balance was achieved.

SUMMARY:
This study aims to evaluate the treatment outcomes of temporomandibular disorders (TMD) using stabilization splints (SS) supported by the T-scan system at Hanoi Medical University Hospital. Thirty-six patients diagnosed with TMD based on the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) received customized stabilization splints. The T-scan system was used to optimize occlusal adjustments by providing real-time digital recordings of occlusal force distribution. Clinical outcomes, including pain intensity (measured by Visual Analog Scale - VAS), maximum comfortable mouth opening (MCO), occlusal time (OT), and disocclusion time (DT), were assessed at baseline, 1 month, and 3 months after treatment. The study investigates the effectiveness of T-scan-assisted occlusal adjustments in improving clinical symptoms and enhancing jaw function in patients with TMD.

DETAILED DESCRIPTION:
This clinical study evaluates the therapeutic effectiveness of stabilization splints (SS) supported by digital occlusal analysis using the T-scan system in patients with temporomandibular disorders (TMD). Thirty-six participants diagnosed with TMD according to the DC/TMD criteria were enrolled and treated at Hanoi Medical University Hospital. Custom-fabricated Michigan-type stabilization splints were provided to all participants. Occlusal adjustments were initially performed using articulating paper and then refined with the T-scan system, which measures occlusal timing and force distribution in real-time.

The primary focus was on improving clinical symptoms such as pain reduction and jaw mobility enhancement. Pain intensity was assessed with the Visual Analog Scale (VAS), and maximum comfortable mouth opening (MCO) was recorded. Occlusal Time (OT) and Disocclusion Time (DT) were evaluated using the T-scan system. Patients were followed up at 1 and 3 months post-treatment to monitor changes.

The study explores the supportive role of digital occlusal adjustment in the conservative management of TMD and highlights the potential of the T-scan system to enhance the precision of splint therapy without direct modification of the natural dentition.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with temporomandibular disorders (TMD) based on the Diagnostic Criteria for Temporomandibular Disorders (DC/TMD).
* Willing and able to wear a stabilization splint as instructed.
* Provided written informed consent.

Exclusion Criteria:

* Presence of systemic diseases (e.g., rheumatoid arthritis, fibromyalgia).
* Unstable general health condition.
* Psychological disorders that could interfere with compliance.
* Ongoing use of other treatments for TMD.
* History of maxillofacial surgery within the past 6 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity (VAS score) | Baseline, 1 month, 3 months
  Pain intensity will be assessed using the Visual Analog Scale (VAS, 0-10) at baseline, 1 month, and 3 months after treatment initiation.

SECONDARY OUTCOMES:
Change in Maximum Comfortable Mouth Opening (MCO) | Baseline, 1 month, 3 months
  Maximum comfortable mouth opening (in millimeters) will be measured between the incisal edges of the upper and lower central incisors at baseline, 1 month, and 3 months.
Change in Occlusal Time (OT) | Baseline, 1 month
  Occlusal Time (in seconds) will be measured by the T-scan system at baseline and after 1 month of splint therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical Univeristy Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No